CLINICAL TRIAL: NCT01021514
Title: Association Between Arterial Wall Uptake of Fluorodeoxyglucose on PET Imaging and sRAGE
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Responsible Party: Korea University Guro Hopital Endocrinology department, Korea University Guro Hospital
Other Study IDs: PET(RAGE)
Record Dates: First submitted 2009-11-27; First posted 2009-11-30 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: sRAGE Level; SUV and TBR Levels in FDG PET
Keywords: sRAGE; SUV; TBR; FDG PET CT; Type 2 DM

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 2 DM, Healthy control: Type 2 DM patients are treating in the Diabetic Clinic of Korea university Guro hospital, and their age- and sex-matched healthy controls are underwent a routine health checkup at Korea university Guro hospital.
- Type 2 DM, Heatlhy control

SUMMARY:
Arteriosclerosis is a dynamic inflammatory disorder. Recently, FDG-PET CT is emerging diagnostic tool of non-invasive technique to detect vulnerable atherosclerotic plaque. And there are arising evidence that sRAGE(soluble Receptor for Advanced glycation End Product) is correlated with metabolic risk. So the investigators will investigate association between sRAGE and FDG-PET uptake in large artery in healthy patient.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis od type 2 DM

Exclusion Criteria:

* Type 1 DM
* Gestational Diabetes
* Severe Liver or Renal disease
* Diagnosis of cancer
* Trauma
* Acute infection or inflammatory disease
* Acute vasculitis or history of vasculitis
* Pregnant or Lactating women
* Dyslipidemia(active state)
* Cardiovascular disease or history of CVD
* Chronic obstructive pulmonary disease
* Any patient by judge of investigator

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: type 2 DM diagnoed according to critereia of American Diabetes Asociation.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2009-01; Primary Completion 2010-08 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyoungmook Choi, MD, PhD, Principal Investigator — Korea University Guro Hospital

REFERENCES:
- [Derived] Yang SJ, Kim S, Hwang SY, Kim TN, Choi HY, Yoo HJ, Seo JA, Kim SG, Kim NH, Baik SH, Choi DS, Choi KM. Association between sRAGE, esRAGE levels and vascular inflammation: analysis with (18)F-fluorodeoxyglucose positron emission tomography. Atherosclerosis. 2012 Feb;220(2):402-6. doi: 10.1016/j.atherosclerosis.2011.11.008. Epub 2011 Nov 16. PMID 22137663